CLINICAL TRIAL: NCT06680349
Title: Two Anti-CD20 Regimens for Fibrillary Glomerulonephritis
Acronym: CD20FG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIBR01
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Fibrillary Glomerulonephritis
Keywords: fibrillary glomerulonephritis; anti-CD20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-CD20 alone (Active Comparator): Lymphoma Protocol consisting of four weekly doses of 375 mg/m2 of rituximab (RTX)
  Interventions: Drug: Anti-CD20 antibodies
- IBCDT (Experimental): Intensive B-cell depletion therapy (IBCDT) which is based on the combination of RTX (given at the dose of 375 mg/m2 every 4 weeks followed by 2 additional doses after 1 and 2 months), CYC (two pulses of 10 mg/kg, corrected according to renal function, on days 4 and 17) and methylprednisolone (three bolus doses of 15 mg/kg) followed by oral prednisone (starting dose 50 mg tapered until complete discontinuation in 4 months).
  Interventions: Drug: Anti-CD20 antibodies

INTERVENTIONS:
Drug: Anti-CD20 antibodies — comparing anti-CD20 (lymphoma protcol, RTX 375 mg/m2 every 4 weeks ) alone Vs. Intensive B-cell depletion therapy (IBCDT) which is based on the combination of RTX (given at the dose of 375 mg/m2 every 4 weeks followed by 2 additional doses after 1 and 2 months), cyclophosphamide (two pulses of 10 mg/kg, corrected according to renal function, on days 4 and 17) and methylprednisolone (three bolus doses of 15 mg/kg) followed by oral prednisone (starting dose 50 mg tapered until complete discontinuation in 4 months).

SUMMARY:
This study aims to evaluate the clinical and histological effects of two rituximab-based regimens in fibrillary glomerulonephritis.

ELIGIBILITY:
Inclusion Criteria:

-Fibrillary glomerulonephritis (biospy proven defined by optical microscopy, immunofluorescence and electron microscopy studies with demonstration of the DNAJB9 protein)

Exclusion Criteria:

* previous treatment with anti-CD20; pregnant; unable to consent. other concomitant GN.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
renal responce | 0, 3 and 6 months
  complete remission (CR), i.e., decrease of proteinuria to <0.5g/day with normal or stable renal function (< 20% increase in serum creatinine); partial remission (PR), i.e., reduction in proteinuria by ≥50% with stable renal function

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni Bosco Hub Hospital, Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No